CLINICAL TRIAL: NCT00734318
Title: A Double Blind, Double Dummy, Randomised, Multicentre, Four Arm Parallel Group Study to Assess the Efficacy and Safety of FlutiForm® pMDI 250/10µg (2 Puffs Bid) vs Fluticasone pMDI 250µg (2 Puffs Bid) Plus Formoterol pMDI 12µg (2 Puffs Bid) Administered Concurrently in Adult Subjects With Severe Persistent, Reversible Asthma.
Brief Title: Study of FlutiForm® Versus Fluticasone Plus Formoterol in Adult Subjects With Severe Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FLT3503; 2007-001633-34
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma, Bronchial
Keywords: Severe asthma; Fluticasone; Formoterol
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Flutiform 250/10 micrograms (Experimental): Flutiform 250/10 micrograms (2 puffs bd)
  Interventions: Drug: Flutiform 250/10 micrograms
- Flutiform 50/5 micrograms (Experimental): Flutiform 50/5 micrograms (2 puffs bd)
  Interventions: Drug: Flutiform 50/5 micrograms
- Flixotide pMDI 250 mcg + foradil pMDI 24 micrograms (Active Comparator): Flixotide pMDI 250 mcg (2 puffs bd) + foradil pMDI 24 50/5 mcg (bd)
  Interventions: Drug: Flixotide pMDI 250 mcg + foradil pMDI 24 micrograms
- Flixotide pMDI 250 micrograms (Active Comparator): Flixatide pMDI 250 micrograms (2 puffs bd)
  Interventions: Drug: Flixotide pMDI 250 micrograms

INTERVENTIONS:
Drug: Flutiform 250/10 micrograms
  Arms: Flutiform 250/10 micrograms
Drug: Flutiform 50/5 micrograms
  Arms: Flutiform 50/5 micrograms
Drug: Flixotide pMDI 250 mcg + foradil pMDI 24 micrograms
  Arms: Flixotide pMDI 250 mcg + foradil pMDI 24 micrograms
Drug: Flixotide pMDI 250 micrograms
  Arms: Flixotide pMDI 250 micrograms

SUMMARY:
The study compares the efficacy and safety of FlutiForm® vs Flixotide® plus Foradil® in the treatment of severe persisent asthma in adult subjects.

DETAILED DESCRIPTION:
This is a study involving a 2 week run-in phase followed by an 8 week double blind treatment phase. During the run-in phase, subjects receive Flixotide®. In the treatment phase subjects will be randomised to one of the four treatment groups and will receive either high dose FlutiForm® and Foradil® plus Flixotide® placebo or low dose FlutiForm® plus Foradil® and Flixotide® placebo or Foradil® plus Flixotide® and FlutiForm® placebo or Flixotide® and FlutiForm® plus Foradil® placebo. Efficacy will be assessed by lung function tests, asthma symptoms, sleep disturbance due to asthma and rescue medication use. Safety will be assessed by adverse events, lab tests, ECGs and vital signs.

ELIGIBILITY:
Inclusion criteria:

1. Male or female subjects at least 18 years old.
2. Females less than one year post-menopausal must have a negative urine pregnancy test recorded at the screening visit prior to the first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner.
3. Known history of severe persistent, reversible asthma for ≥ 6 months prior to the Screening Visit characterised by treatment with ICS at a dose of ≥ 500µg fluticasone or equivalent.
4. Demonstrated a FEV1 of ≥ 40% to ≤ 80% for predicted normal values (Quanjer et al., 1993) during the Screening Visit (Visit 1) and Randomisation Visit (Visit 3) following appropriate withholding of asthma medications (if applicable).

   * No β2-agonist use on day of screening.
   * No use of inhaled combination asthma therapy on day of screening.
   * Inhaled corticosteroids are allowed on day of screening.
5. Documented reversibility of ≥ 15% in FEV1 in the screening phase.
6. Demonstrated satisfactory technique in the use of the study medication.
7. Willing and able to enter information in the electronic diary and attend all study visits.
8. Willing and able to substitute study medication for their pre study prescribed asthma medication for the duration of the study.
9. Written informed consent obtained.

   Inclusion criteria required following run-in:
10. Subject has used rescue medication for at least 3 days AND had at least one night with sleep disturbance (i.e., sleep disturbance score of ≥ 1) OR at least 3 days with asthma symptoms (i.e., a symptom score of ≥ 1) during the last 7 days of the run-in period.

Exclusion criteria:

1. Near fatal or life-threatening (including intubation) asthma within the past year.
2. Hospitalisation or an emergency visit for asthma within the 4 weeks before the screening visit.
3. Known history of systemic (injectable or oral) corticosteroid medication within 1 month of the Screening Visit.
4. Known history of omalizumab use within the past 6 months.
5. Current evidence or known history of any clinically significant disease or abnormality including uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia. 'Clinically significant' is defined as any disease that, in the opinion of the Investigator, would put the subject at risk through study participation, or which would affect the outcome of the study.
6. In the investigator's opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to the Screening Visit.
7. Significant, non-reversible, active pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, tuberculosis).
8. Known Human Immunodeficiency Virus (HIV)-positive status.
9. Subject has a smoking history equivalent to "10 pack years" (i.e., at least 1 pack of 20 cigarettes /day for 10 years or 10 packs/day for 1 year, etc.).
10. Current smoking history within 12 months prior to the Screening Visit.
11. Current evidence or known history of alcohol and/or substance abuse within 12 months prior to the Screening Visit.
12. Subject has taken B-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within the past week.
13. Current use of medications other than those allowed in the protocol that will have an effect on bronchospasm and/or pulmonary function.
14. Current evidence or known history of hypersensitivity or idiosyncratic reaction to test medications or components.
15. Subject has recieved an investigational drug within 30 days of the Screening Visit (12 weeks if an oral or injectable steroid).
16. Subject is currently participating in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1667 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Comparison of FEV1 (Forced expiratory volume in the first second) values. | 8 weeks
  8 weeks on treatment

SECONDARY OUTCOMES:
Other lung function parameters, asthma symptom scores, sleep disturbance due to asthma, rescue medication use, AQLQ, safety assessments. | 8 weeks
  8 week treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Siófok, Hungary

REFERENCES:
- [Derived] Dissanayake S, Jain M, Grothe B, McIver T, Papi A. An evaluation of comparative treatment effects with high and low dose fluticasone propionate/formoterol combination in asthma. Pulm Pharmacol Ther. 2015 Dec;35:19-27. doi: 10.1016/j.pupt.2015.10.001. Epub 2015 Nov 10. PMID 26474679
- [Derived] Bodzenta-Lukaszyk A, Pulka G, Dymek A, Bumbacea D, McIver T, Schwab B, Mansikka H. Efficacy and safety of fluticasone and formoterol in a single pressurized metered dose inhaler. Respir Med. 2011 May;105(5):674-82. doi: 10.1016/j.rmed.2010.11.011. Epub 2010 Dec 31. PMID 21196104
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT3503